CLINICAL TRIAL: NCT05195086
Title: A Pharmacoeconomic Study Comparing the Use of Mycophenolate Mofetil or Cyclophosphamide as Induction Therapy in Lupus Nephritis Patients in Egypt
Status: Completed | Type: Observational
Sponsor: Nada Magdy Mansour (Other)
Responsible Party: Sponsor-Investigator, Nada Magdy Mansour, demonstrator at clinical pharmacy department, Cairo University
Organization: Cairo University (Other)
Other Study IDs: CP3.4.2
Record Dates: First submitted 2022-01-04; First posted 2022-01-18 (Actual); Last update posted 2022-01-18 (Actual); Status verified 2022-01

CONDITIONS: Lupus Nephritis
Keywords: Lupus Nephritis, immunosuppressive agents, Mycophenolic acid, Cyclophosphamide, healthcare costs, cost saving regimen, resource-limited setting, Egypt.
MeSH Terms: conditions — Lupus Nephritis | interventions — Cyclophosphamide; Mycophenolic Acid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes

GROUPS / COHORTS (2):
- Cyc group
  Interventions: Drug: endoxan
- MMF group
  Interventions: Drug: cellcept

INTERVENTIONS:
Drug: endoxan — Immunosuppressant
  Other Names: Cyclophosphamide
  Groups: Cyc group
Drug: cellcept — Immunosuppressant
  Other Names: Mycophenolate Mofetil
  Groups: MMF group

SUMMARY:
The aim of this study is to conduct a pharmacoeconomic analysis to compare the use of Mycophenolate Mofetil or i.v. Cyclophosphamide as induction therapy from a third party payer perspective in LN patients in the Egyptian context

ELIGIBILITY:
Inclusion Criteria:

- LN patients between 18 and 65 years of age who were followed up in the Department of Rheumatology and Rehabilitation were included during the study period. All patients fulfilled at least 4 of the 11 American College of Rheumatology (ACR) revised criteria for the classification of SLE 21. Patients were included if they had active lupus nephritis LN(LN) that was confirmed by Class III, or Class IV, or Class V renal biopsy and which was performed within six months of enrolment. Furthermore, laboratory tests must show active nephritis demonstrated by a clinically significant high level of proteinuria, which might indicate a recent decline in renal function 22. Patients with class III or V LN must have either proteinuria (≥ 2 gm/day) or serum creatinine > 1.3 mg/dl. Patients with class IV must have either proteinuria ≥ 1 gm/day or serum creatinine > 1.3 mg/dl 23. Newly diagnosed patients who were given either IV CYC or oral MMF as induction therapy or patients who needed to be induced when flared up were included in the study.

All patients signed a written informed consent form. For those below the age of 21, written informed consent was obtained from the parents.

Exclusion Criteria:

* Patients were excluded from the study if they had a history of known allergy to study drugs, received previous kidney transplantation, or were on continuous dialysis for more than two weeks before the study. Patients with combinations of membranous and proliferative glomerulonephritis (i.e., class III + V or class IV + V) renal biopsies were not included. Other reasons for exclusion were pregnancy and lactation, pancreatitis, current infection episode requiring IV antibiotics, severe viral infection, history of cancer, or overlapping autoimmune condition.

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Newly diagnosed patients who were given either IV CYC or oral MMF as induction therapy or patients who needed to be induced when flared up were included in the study.
  All patients signed a written informed consent form. For those below the age of 21, written informed consent was obtained from the parents.
Sampling Method: Non-Probability Sample
Enrollment: 122 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2021-06-05 (Actual)

PRIMARY OUTCOMES:
clinical outcomes | 6 months - 12 months
  renal remission
pharmacoeconomic outcomes | 12 months
  comparison of Direct medical costs between both regimens
Quality of life outcomes | baseline and after 12 months
  SF36 Survey comparison between both groups

SECONDARY OUTCOMES:
Adverse events | 12 months
  percentage of adverse events in each group

CONTACTS AND LOCATIONS:
Locations (1):
- Kasr El Aini Hospital, Cairo, Egypt